CLINICAL TRIAL: NCT02588833
Title: A Phase Ib, Open Label, Multiple Ascending Dose, Pilot Study to Assess the Safety, Preliminary Efficacy and Pharmacokinetics of Subcutaneously Administered APL-2 in Subjects With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: Pilot Study to Assess Safety, Preliminary Efficacy and Pharmacokinetics of S.C. Pegcetacoplan (APL-2) in PNH Subjects.
Acronym: PADDOCK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL2-CP-PNH-204
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH; Paroxysmal Nocturnal Hemoglobinuria; Complement inhibitor; Anemia; Hemoglobinuria; Hemolysis; Hematologic diseases; Extravascular hemolysis (EVH); Intravascular hemolysis (IVH); C3 inhibitor
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Anemia; Hemoglobinuria; Hemolysis; Hematologic Diseases | interventions — pegcetacoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): 180 mg pegcetacoplan/day
  Interventions: Drug: Pegcetacoplan
- Cohort 2 (Experimental): 270 mg pegcetacoplan/day
  Interventions: Drug: Pegcetacoplan

INTERVENTIONS:
Drug: Pegcetacoplan — Complement (C3) Inhibitor
  Other Names: APL-2

SUMMARY:
The objectives of the study are to assess the safety, tolerability, preliminary efficacy and PK of multiple subcutaneous (SC) doses of pegcetacoplan in subjects with paroxysmal nocturnal hemoglobinuria (PNH) who have not received treatment with eculizumab in the past.

An exploratory objective of the study is to assess the pharmacodynamics (PD) of multiple SC doses of pegcetacoplan when administered to PNH patients.

DETAILED DESCRIPTION:
This is a Phase Ib, open-label, multiple ascending dose, pilot study in patients with PNH who have not received eculizumab (Soliris)® in the past. Two cohorts of 3 subjects are planned for evaluation.

Safety will be assessed throughout the study; serial blood and urine samples will be collected for these assessments. Blood samples will be collected for the assessment of pegcetacoplan PK. Additional samples for assessment of PD will also be collected.

The study will consist of four parts;

* Part 1: subjects will receive pegcetacoplan for 28 days.
* Part 2A: subjects may continue to receive pegcetacoplan for a further 56 days if there is evidence of perceived clinical benefit following review of available safety, PK and PD data by the investigator and sponsor
* Part 2B/Part 2C: subjects may continue to receive daily pegcetacoplan treatment for up to 364 days if there is ongoing evidence of clinical benefit following review of the available safety, PK and PD data. After completion of Part 2B, subjects could continue treatment with pegcetacoplan by transitioning to an open-label extension study or Part 2C, if enrollment into the extension study was not yet available. Subjects entering Part 2C continued their pegcetacoplan dose and regimen until enrollment in the open-label extension study was available.
* Part 3: Safety follow up Screening will take place within 30 days prior to the start of dosing on Day 1. If needed (see inclusion criteria), Neisseria menigitides types A, C, W, Y and B (administered as two separate vaccinations), Pneumococcal conjugate vaccine or Pneumococcal polysaccharide vaccine 23 (PCV13 or PPSV23, respectively), and Haemophilus influenzae Type B (Hib) vaccinations will be administered at least 14 days prior to dosing on Day 1.

Subjects will be entered into Part 1 of the study on Day 1 at a time designated by the PI. During Part 1, the first 3 daily SC doses of pegcetacoplan (Day 1 to 3) as well as doses on Day 8, 15 and 22 will be administered at the clinical site. From Day 4 to Day 28 daily doses of pegcetacoplan will be administered off-site by a trained study nurse at the subject's home, workplace, or other location convenient to the subject with the exception of those days where dosing is at the clinical site. Following ongoing review of available safety, PK and PD data by the investigator and sponsor, subjects showing evidence of perceived clinical benefit may progress to Part 2A and then to Part 2B of the study and continue to receive daily doses of pegcetacoplan until Day 84 and then until Day 364.

Cohort 2 will not be initiated until all subjects in Cohort 1 have reached the Day 29 visit and the SMC has reviewed emerging safety and efficacy data and determined that, at the initial dose, pegcetacoplan has an acceptable safety and tolerability profile.

The planned length of participation in the study for each subject in Cohort 2 is approximately 444 days (14.5 months) from Day 30 through completion of the Day 414 Exit visit procedures).

The study is planned to take place over approximately 24 months (from screening of Cohort 1 through completion of Cohort 2).

This time period may change in the event that the study is terminated early, additional cohorts are enrolled, additional time is required to review safety between cohorts, or extended safety and PK sampling is added for a cohort.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* At least 18 years old (inclusive)
* Weigh >55 kg and have a body mass index (BMI) ≤38.0 kg/m2
* Diagnosed with PNH (white blood cell (WBC) clone >10%)
* Lactose dehydrogenase (LD) ≥2 times the upper limit of normal
* Last transfusion within 12 months prior to screening
* Platelet count of >30,000/mm3
* Absolute neutrophil count >cells/500 µL
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study
* Males must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study
* Able to provide documentary evidence of Neisseria meningitidis, Pneumococcal conjugate vaccine (multivalent) or Pneumococcal polysaccharide vaccine 23 (PCV13 or PPSV23) and Haemophilus influenzae Type B (Hib) vaccination within 2 years prior to Day 1 dosing, OR willing to receive vaccinations against Neisseria meningitidis at least two weeks prior to dosing on Day 1 with a booster on Day 57, and PCV13 and Hib vaccines at least two weeks prior to dosing on Day 1.
* Willing and able to give informed consent

Exclusion Criteria:

* Prior eculizumab (Soliris)® treatment
* Active bacterial infection
* Known infection with hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* Hereditary complement deficiency
* History of bone marrow transplantation
* Concurrent severe aplastic anemia (SAA), defined as currently receiving immunosuppressive therapy for SAA including but not limited to cyclosporin A, tacrolimus, mycophenolate mofetil or anti-thymocyte globulin.
* Participation in any other investigational drug trial or exposure to another investigational agent, device or procedure within 30 days
* Evidence of QTcF prolongation defined as >450 ms for males and >470 ms for females at screening
* Creatinine clearance (CrCl) <50 mL/min (Cockcroft-Gault formula) at screening
* Breast-feeding women
* History of meningococcal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Grossi, MD, PhD, Study Director — Apellis Pharmaceuticals, Inc.
Locations (7):
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hospital Ampang, Ampang, Selangor, Malaysia
- Waikato Hospital, Hamilton, Waikato Region, New Zealand
- Thailand (3):
  - Ramathibodi Hospital, Bangkok
  - Siriraj hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok

REFERENCES:
- [Derived] Panse J, Daguindau N, Okuyama S, Peffault de Latour R, Schafhausen P, Straetmans N, Al-Adhami M, Persson E, Wong RSM. Improvements in hematologic markers and decreases in fatigue with pegcetacoplan for patients with paroxysmal nocturnal hemoglobinuria and mild or moderate anemia (hemoglobin >/=10 g/dL) who had received eculizumab or were naive to complement inhibitors. PLoS One. 2024 Jul 29;19(7):e0306407. doi: 10.1371/journal.pone.0306407. eCollection 2024. PMID 39079163
- [Derived] Wong RSM, Pullon HWH, Amine I, Bogdanovic A, Deschatelets P, Francois CG, Ignatova K, Issaragrisil S, Niparuck P, Numbenjapon T, Roman E, Sathar J, Xu R, Al-Adhami M, Tan L, Tse E, Grossi FV. Inhibition of C3 with pegcetacoplan results in normalization of hemolysis markers in paroxysmal nocturnal hemoglobinuria. Ann Hematol. 2022 Sep;101(9):1971-1986. doi: 10.1007/s00277-022-04903-x. Epub 2022 Jul 22. PMID 35869170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1b, pilot study was conducted at 9 sites in 5 countries (Hong Kong, Malaysia, New Zealand, Thailand and United States) in subjects with paroxysmal nocturnal hemoglobinuria (PNH) who had not received treatment with eculizumab (Soliris®) in the past, between 01 December 2015 and 26 August 2019. A total of 22 subjects were enrolled.
Pre-assignment Details: Subjects could participate in more than 1 cohort. The study consisted of 3 parts: Part 1 for Cohorts 1 and 2, Part 2 (Part 2A, Part 2B and Part 2C) for Cohort 2 only and Part 3 (safety follow-up). Cohort 2 dosing was not initiated until all subjects in Cohort 1 had completed Part 1 and review of emerging safety and efficacy data. Overall, 2 cohorts of 22 unique subjects were evaluated.
Groups:
- Cohort 1: Subjects received subcutaneous (SC) injections of pegcetacoplan 180 milligrams (mg)/day for up to 28 days.
- Cohort 2: Subjects received SC injections or infusions of pegcetacoplan 270 mg/day for up to 364 days if entering the open-label extension study or, if entering Part 2C, until enrollment in the open-label extension study became available. If clinically indicated on the basis of response, the pegcetacoplan dosage could be increased up to 360 mg/day.
Period: Part 1
Arm/Group | Cohort 1 | Cohort 2
Started | 3 (One subject was enrolled in both cohorts, this subject was enrolled twice.) | 20 (One subject was enrolled in both cohorts, this subject was enrolled twice.)
Completed | 2 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Part 2A
Arm/Group | Cohort 1 | Cohort 2
Started | 0 (Part 2A is not applicable since Cohort 1 subjects proceeded immediately to Part 3.) | 20
Completed | 0 | 18
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Part 2B
Arm/Group | Cohort 1 | Cohort 2
Started | 0 | 18
Completed | 0 | 17
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Part 2C
Arm/Group | Cohort 1 | Cohort 2
Started | 0 | 14 (17 subjects completed Part 2B and 3 entered extension study without participating in Part 2C.)
Completed | 0 | 12
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Part 3 (Safety Follow-up)
Arm/Group | Cohort 1 | Cohort 2
Started | 3 (Only subjects who did not enter extension study or Part 2C entered Part 3.) | 4 (Only subjects who did not enter extension study or Part 2C entered Part 3.)
Completed | 3 | 2
Not Completed | 0 | 2
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat (ITT) population set included all subjects eligible to receive study drug and who received ≥1 dose of study drug. In this study, subjects could participate in more than 1 cohort. Overall, 2 cohorts of 22 unique subjects were evaluated as one subject participated in cohorts 1 and 2.
Groups:
- Cohort 1: Subjects received SC injections of pegcetacoplan 180 mg/day for up to 28 days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 3 | 20 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 19 | 22
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 9 | 10
  Male | 2 | 11 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 1 | 4
  Asian | 0 | 15 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Maori | 0 | 1 | 1
  Other | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 3 | 19 | 22
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs) Including by Severity
Description: TEAEs were defined as adverse events (AEs) that occurred after dosing on Day 1 and up to 30 days after the last dose of study drug. A treatment-related TEAE is defined as a TEAE with a relationship to study drug of probably, possibly, unlikely, or unrelated. A serious adverse event (SAE) is defined as any AE that resulted in death; was life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant incapacity or substantial disruption of ability to conduct normal life functions; was a congenital anomaly or birth defect. TEAEs were graded according to Common Terminology Criteria for Adverse Events v4.03 based on: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death related to AE.
Time Frame: From first dose of study drug (Day 1) up to 30 days after the last dose of study drug, up to approximately 563 days.
Population: The safety population set included all subjects eligible to receive study drug and who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 20
Participants
  All TEAEs | 2 | 18
  Treatment related TEAEs | 2 | 9
  Serious AEs | 1 | 6
  TEAEs leading to study drug discontinuation | 1 | 2
  TEAEs leading to death | 0 | 1
  TEAEs with mild intensity | 0 | 3
  TEAEs with moderate intensity | 2 | 8
  TEAEs with severe intensity | 0 | 5
  TEAEs with life threatening intensity | 0 | 1

2. Primary Outcome: Mean Change From Baseline in Lactate Dehydrogenase (LDH) at Day 365
Description: Serum chemistry assessments of LDH were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the different parts of the treatment period. LDH results were summarized for Cohort 2 only.
Time Frame: Baseline (Day 1) and Day 365.
Population: The ITT population set included all subjects eligible to receive study drug and who received ≥1 dose of study drug. Only subjects analyzed at Day 365 are reported.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
units per liter (U/L) | -2105.2 (1078.79)

3. Primary Outcome: Mean Percentage Change From Baseline in LDH at Day 365
Description: as for outcome 2
Time Frame: Baseline (Day 1) and Day 365.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
percent change | -84.8 (14.04)

4. Primary Outcome: Mean Change From Baseline in Haptoglobin at Day 365
Description: Serum chemistry assessments of haptoglobin were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the different parts of the treatment period. Haptoglobin results were summarized for Cohort 2 only.
Time Frame: Baseline (Day 1) and Day 365.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
gram per liter (g/L) | 0.066 (0.1245)

5. Primary Outcome: Mean Percentage Change From Baseline in Haptoglobin at Day 365
Description: as for outcome 4
Time Frame: Baseline (Day 1) and Day 365.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
percent change | 166.176 (311.3656)

6. Primary Outcome: Mean Change From Baseline in Hemoglobin at Day 365
Description: Hematology assessments of hemoglobin were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the different parts of the treatment period. Hemoglobin results were summarized for Cohort 2 only.
Time Frame: Baseline (Day 1) and Day 365.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
g/L | 3.68 (2.690)

7. Primary Outcome: Mean Percentage Change From Baseline in Hemoglobin at Day 365
Description: as for outcome 6
Time Frame: Baseline (Day 1) and Day 365.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
percent change | 49.86 (43.254)

8. Secondary Outcome: Mean Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Day 365
Description: The FACIT-Fatigue Scale is a 13 item Likert scaled instrument where the subject was presented with 13 statements and asked to indicate their response as it applied to the past 7 days. The 5 possible responses were 'Not at all' (0), 'A little bit (1), 'Somewhat' (2), 'Quite a bit' (3) and 'Very much' (4). There are 13 statements with the total score ranging from 0 to 52 and higher scores indicating better quality of life. The FACIT-Fatigue Scale results were summarized for Cohort 2 only.
Time Frame: Baseline (Day 1) and Day 365.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
score on a scale | 7.1 (11.09)

9. Secondary Outcome: Mean Change From Baseline in Absolute Reticulocyte Count (ARC) at Day 365
Description: Hematology assessments of ARC were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the different parts of the treatment period. ARC results were summarized for Cohort 2 only.
Time Frame: Baseline (Day 1) and Day 365.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
10^9 cells/L | -105.9 (70.28)

10. Secondary Outcome: Mean Percentage Change From Baseline in ARC at Day 365
Description: as for outcome 9
Time Frame: Baseline (Day 1) and Day 365.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
percent change | -47.5 (26.86)

11. Secondary Outcome: Mean Change From Baseline in Total Bilirubin at Day 365
Description: Serum chemistry assessments of total bilirubin were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the 3 parts of the treatment period. Total bilirubin results were summarized for Cohort 2 only.
Time Frame: Baseline (Day 1) and Day 365.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micromole per liter (umol/L)
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
micromole per liter (umol/L) | -29.9 (24.34)

12. Secondary Outcome: Mean Percentage Change From Baseline in Total Bilirubin at Day 365
Description: as for outcome 11
Time Frame: Baseline (Day 1) and Day 365.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
percent change | -60.9 (19.00)

13. Secondary Outcome: Number of Subjects Receiving Red Blood Cell (RBC) Transfusions
Description: The number of on-study RBC transfusions were monitored throughout the treatment period.
Time Frame: From Day 1 up to Day 533.
Population: The ITT population set included all subjects eligible to receive study drug and who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 20
Participants | 1 | 7

ADVERSE EVENTS:
Time Frame: TEAE data is reported from first dose of study drug (Day 1) up to 30 days after the last dose of study drug, up to approximately 563 days.
Description: The safety population set included all subjects eligible to receive study drug and who received ≥1 dose of study drug. One subject was enrolled in both cohorts.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/20
Serious Adverse Events (participants affected / at risk) | 1/3 | 6/20
Other Adverse Events (participants affected / at risk) | 2/3 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=20)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Intravascular haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Paroxysmal nocturnal haemoglobinuria (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=20)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 5 (6)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Hordeolum (Infections and infestations) | 0 (0) | 1 (2)
Nasal abscess (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 1 (4) | 4 (5)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Injection site induration (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 3 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (6)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 2 (4)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (3)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT02588833/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT02588833/SAP_001.pdf